CLINICAL TRIAL: NCT01268501
Title: Clinical Assessment of a New Multifocal Contact Lens With Emmetropic Presbyopes
Brief Title: Clinical Assessment of a Multifocal Contact Lens for People Who Use Reading Glasses Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-319-C-019
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-02

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lotrafilcon B multifocal (Experimental): Lotrafilcon B multifocal contact lenses worn bilaterally for 3 weeks on a daily wear basis
  Interventions: Device: Lotrafilcon B multifocal contact lens

INTERVENTIONS:
Device: Lotrafilcon B multifocal contact lens — Commercially marketed, silicone hydrogel, multifocal, soft contact lenses FDA-approved for up to 4 weeks recommended replacement schedule and up to 6 nights of extended (overnight) wear.
  Other Names: AIR OPTIX® AQUA MULTIFOCAL

SUMMARY:
The purpose of this trial is to evaluate the use of multifocal contact lenses in people who use reading glasses only.

ELIGIBILITY:
Inclusion Criteria:

* Is between 40 and 48 years of age (inclusive).
* Has read and signed the Informed Consent.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Wears reading spectacles for close work.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks of enrollment.
* Evidence of systemic or ocular abnormality, infection, or disease likely to affect successful wear of contact lenses or use of accessory solutions.
* Currently enrolled in a clinical trial.
* Has worn contact lenses previously.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 103 participants were recruited at 25 US sites from December 8, 2010, to January 31, 2011.
Pre-assignment Details: Seven participants were enrolled in the study but not dispensed due to failing inclusion/exclusion criteria (1); withdrawing consent/disinterest (4); discomfort (1); and unacceptable subjective vision (1). These participants are included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Period: Overall Study
Arm/Group | Lotrafilcon B Multifocal
Started | 96
Completed | 87
Not Completed | 9
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — Unacceptable Subjective Vision | 3
Not completed — Handling Difficulties | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lotrafilcon B Multifocal
Number analyzed (Participants) | 96
Age Continuous [Mean (Standard Deviation); unit: years] | 44.9 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Overall Convenience With Contact Lenses
Description: Overall convenience with contact lenses, as interpreted by the participant and reported on a questionnaire as a single, retrospective evaluation of 3 weeks of wear time. Overall convenience is measured on a 4-point scale: 1=very satisfied; 2=satisfied; 3=dissatisfied; 4=very dissatisfied. Results were reported as a percentage of participants who responded, "very satisfied" or "satisfied."
Time Frame: 3 weeks of wear
Population: Per Protocol. Two participants were excluded from analysis due to major protocol deviations as determined by masked review.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lotrafilcon B Multifocal
Number analyzed (Participants) | 85
Percentage of participants | 82.4 [72.6 to 89.8]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 76 days.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Lotrafilcon B Multifocal
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.